CLINICAL TRIAL: NCT01924390
Title: Histological Comparison of Healing Following Tooth Extraction With Ridge Preservation Using Mineralized Freeze Dried Bone Allograft Alone Versus a Combined Mineralized-Demineralized Freeze Dried Bone Allograft
Brief Title: Histological Comparison of Ridge Preservation Using Mineralized FDBA Alone Versus a Combined Mineralized-Demineralized Freeze Dried Bone Allograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Brian L Mealey, Graduate Program Director, Dept of Periodontics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20120278H
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Tooth Extraction
Keywords: Tooth extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mineralized FDBA alone (Active Comparator): Socket grafting with mineralized freeze-dried bone allograft alone
  Interventions: Device: Mineralized freeze-dried bone allograft alone
- Combination of mineralized and deminieralized FDBA (Experimental): Socket grafting with a combination of mineralized and demineralized freeze-dried bone allograft alone
  Interventions: Device: Combination of Mineralized and demineralized freeze-dried bone allograft alone

INTERVENTIONS:
Device: Mineralized freeze-dried bone allograft alone
  Arms: mineralized FDBA alone
Device: Combination of Mineralized and demineralized freeze-dried bone allograft alone
  Arms: Combination of mineralized and deminieralized FDBA

SUMMARY:
This entire protocol involves procedures that are standard care. The purpose of the research is to evaluate whether there are any differences in new bone formation following tooth extraction and grafting of the extraction socket with either 100% mineralized FDBA (FDBA) or a combination of 70% mineralized & 30% demineralized FDBA (DFDBA). Both FDBA and DFDBA are commonly used in dentistry for this purpose. Until recently, there has been no human evidence of differences in new bone formation with one material versus another. Recently, DFDBA has been shown to provide a greater percentage of vital bone formation than FDBA. No studies have been done on materials that provide a combination of demineralized and mineralized FDBA for ridge preservation. That is the purpose of this study.

There will be two subject groups in this study. All subjects will require extraction of at least one non-molar tooth, followed by replacement of the missing teeth with dental implants. Each group will have 22 subjects. The primary distinction between groups will be the use of either a combination of 70% mineralized & 30% demineralized FDBA or 100% mineralized FDBA: Group 1 will have 70% mineralized & 30% demineralized FDBA grafted into the extraction socket for ridge preservation. Group 2 will have 100% mineralized FDBA grafted into the extraction socket for ridge preservation. The allocation of subjects into group 1 or 2 will based on numbers drawn from a stack of sealed envelopes. A small flap will be reflected to an extent about 3-4mm beyond the bony walls of the socket. A measuring stent will be placed and measurements of ridge width and ridge height will be taken and recorded to the nearest 0.5mm. Ridge width will be measured using a ridge caliper at a point approximately 4mm apical to the facial and lingual bony crest. Ridge height will also be measured. The tooth will be extracted and the subject will then be randomized by drawing a sealed envelope from the stack. Either 100% mineralized FDBA or a combination of 70% mineralized & 30% demineralized FDBA will be placed in the socket to restore the ridge to appropriate contour. A dense polytetrafluoroethylene (PTFE) membrane will then be placed over the socket orifice extending about 3mm beyond the bony socket walls. A PTFE suture will be placed over the membrane to secure it in place. Primary closure will not be attempted. The patient will be seen 7-10 days after extraction/ridge preservation to assess healing. The subject will be seen again 21-28 days to remove the PTFE membrane and to assess clinical healing.

At the time of implant placement, the measuring stent and caliper will be used to determine the ridge width and ridge height again. The implant site will be prepared using a hollow trephine which allows retention of the bony core. The bone removed from the osteotomy site remaining in the trephine will be prepared for histologic examination and analyzed for new bone growth. The following histologic parameters will be measured: percent vital bone formation; percent residual graft material; and, percent nonmineralized connective tissue/bone marrow. Following initial preparation of the implant site with the trephine, an implant of the appropriate length and diameter will be placed. A healing abutment will then be placed. All subjects will be examined at 7-10 days following implant placement. The study will end at the time of this follow up visit. The patient will then be referred to his/her restorative dentist for final restoration.

ELIGIBILITY:
Inclusion Criteria:

* single rooted tooth requiring extraction
* have adequate restorative space for a dental implant-retained restoration
* have at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal
* have a dehiscence of the buccal or lingual bony plate of the tooth socket extending no more than 50% of the total depth of the socket

Exclusion Criteria:

* not meeting inclusion criteria
* active localized or systemic infection other than periodontitis.
* inadequate bone dimensions or restorative space dimensions to place a dental implant
* presence of a disease entity, medical condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, or autoimmune diseases.
* positive medical history of endocarditis following oral or dental surgery.
* sensitivity or allergy to Bacitracin, Gentamicin, Polymyxin B Sulfate, alcohol and/or surfactants (per package insert)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at San Antonio (Dental School), San Antonio, Texas, United States

REFERENCES:
- [Background] Eskow AJ, Mealey BL. Evaluation of healing following tooth extraction with ridge preservation using cortical versus cancellous freeze-dried bone allograft. J Periodontol. 2014 Apr;85(4):514-24. doi: 10.1902/jop.2013.130178. Epub 2013 May 31. PMID 23725026
- [Background] Cook DC, Mealey BL. Histologic comparison of healing following tooth extraction with ridge preservation using two different xenograft protocols. J Periodontol. 2013 May;84(5):585-94. doi: 10.1902/jop.2012.120219. Epub 2012 Jun 9. PMID 22680300
- [Background] Wood RA, Mealey BL. Histologic comparison of healing after tooth extraction with ridge preservation using mineralized versus demineralized freeze-dried bone allograft. J Periodontol. 2012 Mar;83(3):329-36. doi: 10.1902/jop.2011.110270. Epub 2011 Jul 12. PMID 21749166
- [Background] Hoang TN, Mealey BL. Histologic comparison of healing after ridge preservation using human demineralized bone matrix putty with one versus two different-sized bone particles. J Periodontol. 2012 Feb;83(2):174-81. doi: 10.1902/jop.2011.110209. Epub 2011 Jun 21. PMID 21692633
- [Background] Beck TM, Mealey BL. Histologic analysis of healing after tooth extraction with ridge preservation using mineralized human bone allograft. J Periodontol. 2010 Dec;81(12):1765-72. doi: 10.1902/jop.2010.100286. Epub 2010 Jul 27. PMID 20653437
- [Derived] Borg TD, Mealey BL. Histologic healing following tooth extraction with ridge preservation using mineralized versus combined mineralized-demineralized freeze-dried bone allograft: a randomized controlled clinical trial. J Periodontol. 2015 Mar;86(3):348-55. doi: 10.1902/jop.2014.140483. Epub 2014 Nov 21. PMID 25415247

RESULTS

PARTICIPANT FLOW:
Groups:
- Mineralized FDBA Alone: Socket grafting with mineralized freeze-dried bone allograft alone
  Mineralized freeze-dried bone allograft alone
- Combination of Mineralized and Demineralized FDBA: Socket grafting with a combination of mineralized and demineralized freeze-dried bone allograft alone
  Combination of Mineralized and demineralized freeze-dried bone allograft alone
Period: Overall Study
Arm/Group | Mineralized FDBA Alone | Combination of Mineralized and Demineralized FDBA
Started | 22 | 22
Completed | 21 | 21
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mineralized FDBA Alone | Combination of Mineralized and Demineralized FDBA | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Full Range); unit: years] | 51 [22 to 78] | 53 [29 to 72] | 52 [22 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent New Vital Bone Formation
Description: Bone core biopsy will be evaluated histologically for percent new vital bone formation
Time Frame: 18-20 weeks
Measure: Mean (Standard Deviation); unit: percentage of vital bone
Arm/Group | Mineralized FDBA Alone | Combination of Mineralized and Demineralized FDBA
Number analyzed (Participants) | 21 | 21
percentage of vital bone | 24.7 (16.0) | 36.2 (11.9)

2. Secondary Outcome: Percent Residual Graft Material and Percent Connective Tissue
Description: Bone core biopsy will be evaluated histologically for percent residual bone graft material and percent connective tissue
Time Frame: 18-20 weeks
Measure: Mean (Standard Deviation); unit: percentage of residual graft
Arm/Group | Mineralized FDBA Alone | Combination of Mineralized and Demineralized FDBA
Number analyzed (Participants) | 21 | 21
percentage of residual graft | 27.0 (13.6) | 18.2 (12.4)

3. Other Pre Specified Outcome: Change in Ridge Width and Ridge Height
Description: Ridge width and height are measured at time of tooth extraction & grafting, and again 18-20 weeks later at time of implant placement. Changes in ridge height and width are determined.
Time Frame: At time of implant placement, which is 18-20 weeks after grafting of extraction socket
Measure: Mean (Standard Deviation); unit: change in ridge width (loss of width mm)
Arm/Group | Mineralized FDBA Alone | Combination of Mineralized and Demineralized FDBA
Number analyzed (Participants) | 21 | 21
change in ridge width (loss of width mm) | 1.63 (1.18) | 1.19 (1.36)

ADVERSE EVENTS:
Arm/Group | Mineralized FDBA Alone | Combination of Mineralized and Demineralized FDBA
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No